CLINICAL TRIAL: NCT00435864
Title: Pilot, Multicenter and Prospective Study of the Natural Killer Index From Hematopoietic Stem Cell Graft at a Genotypic, Phenotypic and Functional Level
Brief Title: Natural Killer Index From Hematopoietic Stem Cell Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BRD 06/6-N; ID RCB 2007-A00002-51
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloblastic Leukemia; Chronic Myeloid Leukemia
Keywords: recipient of a HSC graft in Acute Myeloblastic Leukemia therapy; recipient of a HSC graft in others pathologies treated in hematology of Nantes university hospital or Angers university hospital; donors are healthy subjects
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- allogeneic donor from a file (Other)
  Interventions: Procedure: Blood test
- Registry geno-identical donor family (Other)
  Interventions: Procedure: Blood test
- transplantation of HSCs derived from placental blood (Other)
  Interventions: Procedure: Blood test

INTERVENTIONS:
Procedure: Blood test — The study of KIR and HLA genes will be performed on samples of cord blood or peripheral blood donor and recipient before transplant For grafts from placental cord blood, we do ask any additional samples.

SUMMARY:
Numerous studies about the potential role of NK alloreactive during a n hematopoietic stem cells graft are based on genotypical analyses of the KIR receptors and on genotypic incompatibilities between KIR and HLA for couple donor/recipient. There is still a lot of issues non resolved: Are KIR really expressed and how occur their expression during time when hematopoietic reconstitution? Is it depending on HLA of the recipient?If KIR are expressed, what are the mechanisms of alloreactivity of NK cells? Are NK able to lyse tumoral cells? Could alloreactive NK cells constitute a therapeutic tool able to induce tolerance and elimination of leukemia during hematopoietic stem cells grafts?

ELIGIBILITY:
Inclusion Criteria:

* Age superior to 1 year
* Patient that will be treated by an HSC graft
* Initial pathology of recipient: acute lymphoblastic leukemia, acute myeloblastic leukemia, chronic myeloid leukemia

Exclusion Criteria:

* Patient already included in a study with an exclusion period
* HIV + or HCV + serology during pre-graft analysis
* Patient already treated by an allograft of HSC

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Estimate in the pilot study the percentage of different NK cell populations during hematopoietic reconstitution after HSCT with regard to the KIR and HLA genotypes of donor / recipient | J60 post-HSCT

SECONDARY OUTCOMES:
Genetic analysis of KIR and HLA incompatibility of donor and recipient - Rate of in vitro amplification of NK cells from the donor - Assess the percentage of NK cells from the donor | J60 post-HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Mechinaud, md, Principal Investigator — Nantes University Hospital; Patrice Chevallier, MD, Principal Investigator — Nantes University Hospital; Nadège Corradini, MD, Principal Investigator — Nantes University Hospital; Norbert Ifrah, MD, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU de Nantes, Nantes, France